CLINICAL TRIAL: NCT03976336
Title: Evaluating the Tolerability and Effects of Berberine on Major Metabolic Biomarkers: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, James Backes, PharmD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00143015
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Berberine (Experimental)
  Interventions: Dietary Supplement: Berberine
- Identical Placebo (Placebo Comparator)
  Interventions: Other: Identical Placebo

INTERVENTIONS:
Dietary Supplement: Berberine — 500 mg berberine (1 capsule) with breakfast and 1000 mg (2 capsules) with the evening meal, 1500 mg total
  Arms: Berberine
Other: Identical Placebo — 500 mg (1 capsule) with breakfast and 1000 mg (2 capsules) with the evening meal, 1500 mg total
  Arms: Identical Placebo

SUMMARY:
Berberine is a dietary supplement that comes from the roots, stems, and bark of various plants and has been used for centuries in traditional Chinese medicine. It may help lower cholesterol, lower blood sugar, and reduce inflammation.Very few studies have been done in the United States to show how berberine effects cholesterol and blood sugar. This study is looking to see how berberine changes cholesterol and blood sugar, and to see how well it is tolerated.Berberine is not a prescription medication but it appears to have similar actions to common prescription medications to lower cholesterol like statins, and to lower blood sugar like metformin. We are studying berberine to see if it may be a good option for people that do not want to take prescription medications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and older
* Current LDL-C of ≥80 mg/dL or higher
* Current fasting triglyceride level of ≥300 mg/dL
* Meets current criteria for metabolic syndrome (≥3 of the following):

Waist circumference ≥ 35" female or ≥40" for male:

Triglycerides ≥ 150 mg/dL:

Low HDL-c <40 mg/dL male or <50 mg/dL female:

Elevated blood pressure ≥ 130/85 mmHg (or on BP medication):

Elevated fasting blood glucose ≥100 mg/dL

* A male or a non-pregnant female
* Mentally competent to understand study rationale and protocol
* Able to speak and read English

Exclusion Criteria:

* Currently taking any lipid-altering agents including but not limited to statins, niacin (>500 mg), bile-acid sequestrants, ezetimibe, fibrates, and Omega-3 fish/krill oils (>1000 mg EPA/DHA).
* Prior evidence of a vascular event (e.g. stroke, myocardial infarction, revascularization, peripheral vascular disease)
* Current use of any oral hypoglycemia agent or parenteral medication for diabetes mellitus (e.g. GLP-1 agonists, insulin)
* Currently taking any drugs with the potential to interact with berberine, including but not limited to cyclosporine, simvastatin, lovastatin, metformin, saquinavir, darunavir, tacrolimus, sirolimus.
* Previous history of diabetes mellitus, HbA1c ≥ 6.5%, or FPG > 126 mg/dL
* Chronic disease involving, hepatic, renal, or coronary heart disease, systemic infection (e.g. HIV) or organ transplantation
* Currently taking systemic steroidal drugs
* Dependence on alcohol (> 10 drinks per week) or illicit drugs
* Pregnant or lactating
* Participation in any other clinical trial within the last 30 days
* Presence of any medical or psychological condition that in the opinion of the investigator will compromise safe subject participation for the duration of the study
* Acute or chronic GI conditions (e.g. irritable bowel syndrome, ulcerative colitis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in LDL Cholesterol | Baseline to week 12
  LDL cholesterol measured by fasting blood sample
Change in Hemoglobin A1c | Baseline to week 12
  Glucose control as measured by fasting blood sample

SECONDARY OUTCOMES:
Number of participants with adverse events | Week 4, Week 8, and Week 12
  Number of participants with adverse events will be measured by a monthly follow-up questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James Backes, PharmD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No